CLINICAL TRIAL: NCT07376876
Title: Indocyanine Green-guided Omental Shield Anastomosis (ICG-OSA) for Cervical Esophagogastric Anastomosis in Minimally Invasive McKeown Esophagectomy: a Single-center, Single-arm, Open-label Clinical Study
Brief Title: Indocyanine Green-guided Omental Shield Anastomosis for Cervical Esophagogastric Anastomosis in Minimally Invasive McKeown Esophagectomy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, WEI GUO, director, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICG-OSA for anastomosis; 0 (Other: Army Medical Center , Army Medical University)
Record Dates: First submitted 2026-01-02; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC); Esophageal Cancer
Keywords: Indocyanine Green Fluorescence Navigation; Anastomotic Leakage; Omental Shield; Esophageal Squamous Cell Carcinoma (ESCC)
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Intervention Model Description: Step 1: ICG-Guided Gastric Conduit Prep: IV ICG , fluorescence laparoscopy assesses gastroepiploic arcade (Koskas types) and perfusion zones (red=good, blue=poor), marks optimal anastomotic site on greater curvature, optimizes conduit tailoring. Step 2: T-Shaped Stapled Anastomosis: 1cm opening on posterior greater curvature wall at best perfusion zone, side-to-side stapling of posterior esophagus to greater curvature, closes common opening, reinforces with absorbable sutures. Step 3: Omental Shield: mobilizes pedicled omentum with good blood supply, 360° sleeve-wrap of anastomosis + 2cm area, fixes with 4-6 absorbable sutures to gastric wall above/below, ensures no tension/torsion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Indocyanine Green-Guided Omental Shield Anastomosis (ICG-OSA) Intervention Group (Experimental)
  Interventions: Procedure: Indocyanine green-guided omental shield anastomosis for cervical esophagogastric anastomosis

INTERVENTIONS:
Procedure: Indocyanine green-guided omental shield anastomosis for cervical esophagogastric anastomosis — Step 1: ICG-guided gastric conduit prep: IV ICG fluorescence laparoscopy assesses gastroepiploic arcade (Koskas types) and perfusion zones (red=good, blue=poor), marks optimal anastomotic site on greater curvature, optimizes conduit tailoring. Step 2: T-Shaped Stapled Anastomosis**: 1cm opening on posterior greater curvature wall at best perfusion zone, side-to-side stapling of posterior esophagus to greater curvature, closes common opening, reinforces with absorbable sutures. Step 3: Omental Shield: mobilizes pedicled omentum with good blood supply, 360° sleeve-wrap of anastomosis + 2cm area, fixes with 4-6 absorbable sutures to gastric wall above/below, ensures no tension/torsion.

SUMMARY:
Brief Summary Study title: Indocyanine green (ICG)-guided omental shield anastomosis (ICG-OSA) technique for cervical esophagogastric anastomosis in esophageal cancer surgery Purpose: To evaluate whether a novel surgical technique can reduce the risk of anastomotic leakage after minimally invasive esophageal cancer surgery.

Eligible participants: Adults aged 18-80 years with histologically confirmed esophageal squamous cell carcinoma (ESCC) in the middle or lower thoracic esophagus who are scheduled for esophagectomy.

The technique: All participants will undergo the ICG-OSA procedure, which uses indocyanine green fluorescence imaging to assess gastric perfusion, creates a T-shaped esophagogastric anastomosis, and wraps the anastomosis with a pedicled omental flap.

Outcome assessments: The primary outcome is anastomotic leakage rate within 30 days after surgery. Secondary assessments include surgical site infection, anastomotic stricture, and hospitalization costs.

Study site: Daping Hospital, Army Medical Center, Chongqing, China Study duration: December 2025 to March 2027 Contact: For more information, please contact the research team at Daping hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 80 years, of both sexes;
2. Pathological diagnosis: Histologically confirmed esophageal squamous cell carcinoma (ESCC) by biopsy;
3. Clinical staging: Preoperative clinical stage cT1-4aN0-3M0 (according to the 8th edition AJCC staging criteria), evaluated by the thoracic surgery team as eligible for radical McKeown esophagectomy;
4. Performance status ECOG 0-1；
5. Major organ function (cardiovascular, respiratory, digestive, hematological systems) assessed as having no contraindications for chemotherapy or immunotherapy, and no surgical contraindications;
6. Able to understand and comply with study protocol requirements, and willing to accept and undergo standardized postoperative follow-up;
7. Able to understand and sign the informed consent form.

Exclusion Criteria:

1. Allergy history: History of allergy to indocyanine green (ICG), iodide, or iodinated contrast agents (ICG contains iodine, and allergy may cause severe anaphylactic reactions);
2. Severe hepatic or renal dysfunction: Severe hepatic insufficiency (Child-Pugh Class C) or severe renal insufficiency (eGFR <30 mL/min/1.73 m²), affecting ICG metabolism and excretion;
3. Unfavorable tumor location: Tumor located in the cervical or upper thoracic esophagus (<25 cm from the incisors), making it difficult to ensure negative proximal resection margin;
4. Previous surgery history: Prior history of esophageal, gastric, or mediastinal surgery resulting in altered anatomy or severe adhesions;
5. Multiple primary cancers: Concurrent active malignant tumors in other sites (except cured basal cell carcinoma of the skin or cervical carcinoma in situ);
6. Special physiological status: Pregnant or lactating women, or those with planned pregnancy during the study period who are unwilling to use effective contraception;
7. Cognitive and behavioral issues: Presence of severe psychiatric illness, cognitive impairment, or history of substance abuse that would preclude compliance with study procedures;
8. Participation in other studies: Currently enrolled in other interventional clinical trials that may interfere with the results of this study;
9. Investigator judgment: Investigator considers the patient unsuitable for this clinical study (e.g., intraoperative exploration reveals severe tumor invasion of major structures such as the aorta or trachea, making R0 resection unachievable).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leakage rate within 30 days postoperatively | Up to 30 days postoperatively (critical assessment window: postoperative day 7±1）
  Anastomotic leakage rate assessed by clinical evaluation, computed tomography (CT) scan with oral contrast, and endoscopy according to ECCG criteria.

SECONDARY OUTCOMES:
Subclinical anastomotic leakage rate | Daily through postoperative day 30
  Turbid mediastinal drainage fluid with positive bacterial culture, but requiring no intervention (i.e., no puncture drainage, stent placement, or surgery); daily recording of drainage fluid characteristics, with positive culture results confirmed by laboratory reports.
Postoperative anastomotic stenosis rate | 6 months postoperatively
  Anastomotic stricture rate diagnosed by endoscopy and dysphagia symptoms.
Anastomotic leakage-related complication rate | Up to 30 days postoperatively
  Complications directly related to anastomotic leakage, including pulmonary infection, empyema, mediastinal infection, and sepsis. Complications will be graded using the Clavien-Dindo classification system. Diagnosis will be confirmed by clinical symptoms (fever, leukocytosis), microbiological cultures, and imaging findings (CT scan showing fluid collections or air-fluid levels). Each complication will be documented with onset date, severity grade, and required interventions.
Health economic indicators | From hospital admission through hospital discharge, an average of 10 days
  Total medical costs from hospital admission to discharge, including operation fees, anesthesia, medication, laboratory tests, imaging studies, hospital bed, and other related expenses. Data will be extracted from the hospital information system (HIS) at discharge and recorded in the case report form.Number of days from the date of surgery to hospital discharge, calculated as (discharge date minus surgery date + 1 day).

OTHER OUTCOMES:
Technique-related adverse events | From intraoperative period through 30 days postoperatively
  1. ICG-related reactions: Allergic reactions (rash, anaphylaxis).
  2. Gastric conduit complications: Ischemia/necrosis of gastric tube, gastric emptying disorder, staple line bleeding.
  3. Omental flap complications: Omental necrosis, poor wound healing at omental harvest site.
  4. Anastomotic technical issues: Stapler misfire, anastomotic bleeding requiring intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Army Medical Center of the People's Liberation Army, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol and Statistical Analysis Plan (2025-12-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT07376876/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Study Protocol and Statistical Analysis Plan V2 (2025-12-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT07376876/Prot_SAP_001.pdf